CLINICAL TRIAL: NCT06747585
Title: A Phase I/II, Open-Label, Multicenter Study of ALE.P02 (Claudin-1 Targeted Antibody-Drug Conjugate) as a Monotherapy in Adult Patients With Selected Advanced or Metastatic CLDN1+Squamous Solid Tumors
Brief Title: A Study to Investigate ALE.P02 as Monotherapy in Adult Patients With Selected CLDN1+ Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alentis Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALE.P02.01; 2024-515459-39-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-17; First posted 2024-12-24 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-10

CONDITIONS: Squamous Non-small-cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; Cervical Squamous Cell Carcinoma; Esophageal Squamous Cell Carcinoma
Keywords: Claudin-1 Targeted Antibody-Drug Conjugate; Monotherapy; First-in-Human; Recommended Phase 2 dose; Recommended dose for expansion
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I Dose Escalation- ALE.P02 (Experimental): Patients will receive ALE.P02 as monotherapy via intravenous infusion. The ALE.P02 will be given at an escalated dose until Maximum tolerated dose (MTD) and/or a safe recommended Dose for Expansion (RDE) is determined in Phase I dose escalation part of the study.
  Interventions: Drug: ALE.P02
- Phase I Dose Expansion- ALE.P02 (Experimental): Patients will receive ALE.P02 as monotherapy via intravenous infusion. The safe recommended dose of ALE.P02 will be given in Phase I dose expansion part of the study to identify Recommended Phase II Dose (RP2D) for Phase II.
  Interventions: Drug: ALE.P02
- Phase II- ALE.P02 (Experimental): Patients will receive ALE.P02 as monotherapy via intravenous infusion at the RP2D, or according to the dosing schedule after the dose expansion phase.
  Interventions: Drug: ALE.P02

INTERVENTIONS:
Drug: ALE.P02 — ALE.P02, will be administered by IV infusion according to the assigned arms.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic, pharmacodynamic, preliminary anti-tumor activity, and to determine the recommended Phase II dose (RP2D) of the ALE.P02 monotherapy in adult patients with selected squamous solid tumors.

DETAILED DESCRIPTION:
This Study has a Phase I ALE.P02 monotherapy dose escalation and recommended dose for expansion (RDE) study and a Phase II study of ALE.P02 as monotherapy at RP2D in adult patients with selected advanced or metastatic Claudin-1 positive (CLDN1+) cancers.

ELIGIBILITY:
Inclusion Criteria:

* Have disease and treatment history as: Have histologically or cytologically confirmed advanced locally recurrent and inoperable or metastatic SqNSCLC, HNSCC (nasopharyngeal cancer included), ESCC or CSCC.
* Phase I Dose Escalation: Have received at least one systemic standard of care regimen and being refractory or intolerant to the treatment.
* Phase I RDE and Phase II: Have received no more than 2 lines of systemic standard of care regimen and being refractory or intolerant to the treatment.
* Have provided tissue for CLDN1 analysis in a central laboratory.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group Performance Scale.
* Demonstrate adequate bone marrow and organ function.
* Patients must have recovered from all toxicities led by prior treatment.
* Have measurable disease based on RECIST 1.1 as determined by the site.

Exclusion Criteria:

* Diagnosed with cancers of predominantly non-squamous histology (eg, adenosquamous carcinoma) or adenocarcinoma.
* Has received antineoplastic therapies prior to study intervention within specified time frame.
* Has rapidly progressing disease (eg, tumor bleeding, uncontrolled tumor pain).
* Patients with uncontrolled diabetes.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has clinically significant gastrointestinal bleeding and has an active infection requiring systemic treatment and has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the clinical study, interfere with the patient's participation for the full duration of the clinical study, or is not in the best interest of the patient to participate.
* Concomitant use of drugs that are known to prolong or shorten QT and/or have known risk of Torsades de Pointes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2028-02-15 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicities (DLTs) | Up to 28 days
  DLTs as defines in the protocol will be assessed to evaluate safety and tolerability of ALE.P02 (Phase I Dose Escalation), and to establish RP2D for ALE.P02 (Phase I RDE).
Number of Patients with Adverse Events | Screening (day -28 to day -1) up to Safety follow-up (30 ± 5 days post last dose [Up to 3.5 years])
  Adverse events will be assessed to evaluate safety and tolerability of ALE.P02 (Phase I Dose Escalation), and to establish RP2D for ALE.P02 (Phase I RDE).
Overall Response Rate (ORR) (Phase I) | From ALE.P02 treatment initiation until at or prior to initiation of the use of new anti-cancer therapy (Up to 3.5 years)
  The ORR is the proportion of patients with a best overall response (BOR) of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1.) This is assessed to establish RP2D for ALE.P02 (Phase I RDE)
Duration of Response (DoR) (Phase I) | From ALE.P02 treatment initiation until disease progression or study completion (Up to 3.5 years)
  The DoR is defined for patients achieving a confirmed CR or PR as the time from the initial response of CR or PR per Investigator review according to RECIST 1.1 to disease progression or death of any cause, whichever occurs earlier. This is assessed to establish RP2D for ALE.P02 (Phase I RDE).
Overall Response Rate (ORR) (Phase II) | From ALE.P02 treatment initiation until at or prior to initiation of the use of new anti-cancer therapy (Up to 3.5 years)
  The ORR is assessed to assess anti-tumor activity of ALE.P02 (Phase II).
Duration of Response (DoR) (Phase II) | From ALE.P02 treatment initiation until disease progression or study completion (Up to 3.5 years)
  The DoR is assessed to assess anti-tumor activity of ALE.P02 (Phase II).

SECONDARY OUTCOMES:
Disease control rate (DCR) (Phase I and II) | From ALE.P02 treatment initiation until at or prior to initiation of the use of new anti-cancer therapy (Up to 3.5 years)
  The DCR is defined as the proportion of patients with a confirmed BOR of CR or PR or stable disease (SD) per Investigator review according to RECIST 1.1 at or prior to initiation of the use of new anti-cancer therapy. This is assessed to evaluate preliminary evidence of anti-tumor activity of ALE.P02 (Phase I and II).
Median Progression-Free Survival (PFS) at 6 and 12 Months (Phase I and II) | At 6 and 12 months after initiation of ALE.P02 treatment
  The PFS is defined as time from first study treatment to a documented disease progression according to RECIST 1.1, as determined by the Investigator, or death due to any cause, whichever occurs earlier. This is assessed to evaluate preliminary evidence of anti-tumor activity of ALE.P02 (Phase I and II).
Median Overall Survival (OS) at 6, 12, and 24 Months (Phase I and II) | At 6, 12, and 24 months after initiation of ALE.P02 treatment
  The OS is defined as time from first study treatment to death due to any cause. This is assessed to evaluate preliminary evidence of anti-tumor activity of ALE.P02 (Phase I and II).
Blood Concentration of ALE.P02 Antibody-drug Conjugate (ADC) | Phase I and II: Cycle 1 Day 1 until at end of treatment visit (EoT) (Up to 3.5 years)
  Concentrations of ALE.P02 ADC in blood will be measured at each scheduled time point per arms to assess the pharmacokinetic (PK) profile of ALE.P02.
Blood Concentration of Total Antibody | Phase I and II: Cycle 1 Day 1 until at EoT (Up to 3.5 years)
  Total antibody in blood will be measured at each scheduled time point per arms to assess the PK profile of ALE.P02.
Blood Concentrations of Payload | Phase I and II: Cycle 1 Day 1 until at EoT (Up to 3.5 years)
  Concentrations of payload in blood will be measured at each scheduled time point per arms to assess the PK profile of ALE.P02.
Area under the concentration-time curve over the dosing interval (AUCtau) | Phase I and II: Cycle 1 Day 1 until at EoT (Up to 3.5 years)
  The AUCtau of ALE.P02 will be measured to assess the pharmacokinetic (PK) profile of ALE.P02.
Area under the concentration-time curve from pre-dose (time 0) to the time of the last quantifiable concentration (AUClast) | Phase I and II: Cycle 1 Day 1 until at EoT (Up to 3.5 years)
  The AUClast of ALE.P02 will be measured to assess the PK profile of ALE.P02.
Area under the concentration-time curve from pre-dose (time 0) extrapolated to infinite time (AUCinf) | Phase I and II: Cycle 1 Day 1 until at EoT (Up to 3.5 years)
  The AUCinf of ALE.P02 will be measured to assess the PK profile of ALE.P02.
Maximum Concentration (Cmax) | Phase I and II: Cycle 1 Day 1 until at EoT (Up to 3.5 years)
  The Cmax of ALE.P02 will be measured to assess the PK profile of ALE.P02. It is determined directly from the concentration-time profile.
Minimum concentration (Cmin) | Phase I and II: Cycle 1 Day 1 until at EoT (Up to 3.5 years)
  The Cmin of ALE.P02 will be measured to assess the PK profile of ALE.P02. It is determined directly from the concentration-time profile.
Concentration at the end of a Dosing Interval (Ctrough) | Phase I and II: Cycle 1 Day 1 until at EoT (Up to 3.5 years)
  The Ctrough of ALE.P02 will be measured to assess the PK profile of ALE.P02.
The terminal elimination rate constant (KeL) | Phase I and II: Cycle 1 Day 1 until at EoT (Up to 3.5 years)
  The KeL of ALE.P02 will be measured to assess the PK profile of ALE.P02. It is determined by selection of at least three data points on the terminal phase of the concentration-time curve.
Terminal elimination half-life (t½) | Phase I and II: Cycle 1 Day 1 until at EoT (Up to 3.5 years)
  The t½ of ALE.P02 will be measured to assess the PK profile of ALE.P02.
Time of Maximum Concentration (tmax) | Phase I and II: Cycle 1 Day 1 until at EoT (Up to 3.5 years)
  The tmax of ALE.P02 will be measured to assess the PK profile of ALE.P02.
Average Concentration (Cavg) | Phase I and II: Cycle 1 Day 1 until at EoT (Up to 3.5 years)
  The Cavg of ALE.P02 will be measured to assess the PK profile of ALE.P02.
Number of Patients with Presence of anti-ALE.P02 Antibodies | Phase I and II: Cycle 1 Day 1 until at EoT (Up to 3.5 years)
  Presence of anti-ALE.P02 Antibodies will be assessed to evaluate the immunogenicity of ALE.P02.

CONTACTS AND LOCATIONS:
Locations (32):
- United States (8):
  - Mayo Foundation for Medical Education and Research - Mayo Cl, Scottsdale, Arizona
  - Providence Medical Foundation, Fullerton, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - The University of Chicago Medical Center - Oncology, Chicago, Illinois
  - Norton Cancer Institue Downtown, Louisville, Kentucky
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NEXT Oncology Virginia, Fairfax, Virginia
- France (3):
  - Institut Bergonie, Bordeaux
  - CHRU De Lille- Hôpital Claude Huriez - Medical Oncology, Lille
  - Institut Gustave Roussy, Villejuif
- Chinese University of Hong Kong - Prince of Wales Hospital, Shatin, N.T., Hong Kong
- Italy (5):
  - Ospedale San Raffaele, IRCCS, Milan
  - IEO - Istituto Europeo di Oncologia, IRCCS, Milan
  - Ospedale Santa Maria delle Croci di Ravenna Oncologia, Ravenna
  - PU A. Gemelli, Universita Cattolica del Sacro Cuore, Roma
  - Centro Ricerche Cliniche Verona, Verona
- Singapore (2):
  - National University Cancer Institue, Singapore, South West
  - National Cancer Centre Singapore, Singapore, South West
- South Korea (3):
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (7):
  - START Madrid- Centro Integral Oncologico Clara Campal, PAU de Sanchinarro, Madrid
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - NEXT Oncology Barcelona, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - START Hospital HM Nou Delfos, Barcelona
  - Hospital Universitario Virgen De La Victoria, Málaga
  - Hospital Universitario Y Politécnico La Fe, Valencia
- Taiwan (3):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - National Taiwan University Hospital, Taipei
  - Buddihist Tzu Chi Medical Foundation - Taipei Tzu Chi Hospital, Taipei